CLINICAL TRIAL: NCT02615002
Title: Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose Ranging Study of Piromelatine in Patients With Mild Dementia Due to Alzheimer's Disease
Brief Title: Safety and Efficacy of Piromelatine in Mild Alzheimer's Disease Patients (ReCOGNITION)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuP11-AD2
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease
Keywords: Cognition; mild Alzheimer's disease; Sleep
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(2-(5-methoxy-indol-3-yl)-ethyl)-4-oxo-4H-pyran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Piromelatine 5 mg (Experimental): 2 weeks of Placebo (run-in), followed by 26 weeks of 5 mg tablets once daily.
  Interventions: Drug: Piromelatine
- Piromelatine 20 mg (Experimental): 2 weeks of Placebo (run-in), followed by 26 weeks of 20 mg tablets once daily.
  Interventions: Drug: Piromelatine
- Piromelatine 50 mg (Experimental): 2 weeks of Placebo (run-in), followed by 26 weeks of 50 mg tablets once daily.
  Interventions: Drug: Piromelatine
- Placebo (Placebo Comparator): 2 weeks of Placebo (run-in), followed by 26 weeks of Placebo tablets once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piromelatine
  Other Names: Neu-P11
  Arms: Piromelatine 20 mg; Piromelatine 5 mg; Piromelatine 50 mg
Drug: Placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
This study is a Phase 2, randomized, placebo-controlled, dose-ranging study of piromelatine (5, 20, and 50 mg daily for 6 months) versus placebo to determine an effective dose based on efficacy (cognitive performance), safety, and tolerability in patients with mild dementia due to Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Patients with a documented history of mild dementia due to AD for at least 6 months, having a Mini-Mental State Examination (MMSE) score of 20 to 27 (inclusive) at Screening.

A score of 27 is allowed only if accompanied by a score of ≥ 12 in the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-cog) ADAS-cog11 portion of the ADAS-cog14 at screening, and a Clinical Dementia Rating Global Score (CDR-GS) of 0.5 or 1 will be recruited and further screened for eligibility. Caregiver commitment to the study is also necessary.

At Screening (Visit 1), patients will undergo neuropsychiatric assessments, psychometric testing, and general medical assessments (including medical history, pre-existing conditions, physical examination, vital signs, and ECG). If patients have not had brain imaging with findings consistent with the diagnosis of dementia due to AD in the last 12 months, a computed tomography (CT) or magnetic resonance imaging (MRI) scan will be obtained to rule out clinically significant comorbid pathologies.

Eligible patients will start a 2-week run-in period of placebo (single-blind), followed by 26 weeks of double-blind treatment comprising administration of piromelatine or placebo, for a total treatment duration of 28 weeks. During the double-blind period, patients will be enrolled in a 1.2:1:1:1 randomization ratio to the 4 trial arms (placebo [1.2], and the equal piromelatine treatment arms 5, 20, and 50 mg [1:1:1]).

Intermediate visits will be carried out at 4 weeks (Visit 3) and 13 weeks (Visit 4) after randomization. A follow-up phone call to elicit any safety concerns will be completed 2 weeks after the last dose of study medication. Patients who discontinue before Visit 5 (Week 26) will be brought back for a termination visit.

Assuming an effect size between the treatment dose and placebo of 0.35 over 26 weeks, a significant level (α) of 0.05, and power of 88%, a sample size of 143 patients for the placebo arm and 119 patients for each of the 3 piromelatine arms is calculated. Assuming a 50% screen failure rate and allowing for 15% patient withdrawal, 1150 patients should be screened to randomly assign 575 patients, of whom it is expected that 500 will complete the study.

Piromelatine (5, 20, and 50 mg tablets) and placebo will be administered orally, once daily after a meal, before habitual bedtime, preferably between 2100h and 2300h. Patients will be required to spend at least 2 hours a day exposed to daylight.

ELIGIBILITY:
Inclusion Criteria:

* Patient and caregiver are willing to take part in the entire study
* Signed informed consent from the patient and the caregiver
* Patient has a documented history either in medical records or from an informant of cognitive decline over at least 6 months
* Patient has mild probable AD as consistent with criteria established by the National Institute on Aging and Alzheimer's Association (NIA-AA).
* CT/MRI scan with finding consisting of probable AD obtained during the last 12 months before Screening
* Patient has an MMSE score of 21-26 (inclusive) at Screening
* Patient has a Clinical Dementia Rating Global Score (CDR-GS) of 0.5-1 (mild dementia) at Screening
* Patients receiving prescribed drugs for treatment of AD including acetyl cholinesterase inhibitors [eg, donepezil, galantamine, rivastigmine] should be on a stable dose for at least 3 months before Screening
* Patient has a negative drug screen (benzodiazepines or opiates) at Screening
* Female patients must have had last natural menstruation ≥ 24 months before Screening, OR being surgically sterile
* Male patients must agree to the use of effective contraception if the female partner is of childbearing potential, OR be surgically sterile

Exclusion Criteria:

* Patient has an alternative cause for dementia other than AD as determined by CT or MRI scan
* Patient has evidence of any clinically significant neurodegenerative disease
* Patient has been diagnosed with the following Axis I disorders (DSM V criteria)
* Patient has a history of uncontrolled or untreated cardiovascular, endocrine, gastrointestinal, respiratory, or rheumatologic disorders within the past 5 years
* Patient has severe pain that is likely to interfere with sleep
* Continuous use of benzodiazepines or other sedative-hypnotics during the 2 weeks before Screening
* Use of any kind of melatonin/melatonin agonist during the 2 weeks before Screening
* Patient has known or suspected hypersensitivity to exogenous melatonin or melatonin receptor agonists
* Patients with an irregular lifestyle or life pattern (eg, shift workers, patients likely to be jet lagged).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-11; Primary Completion 2019-06 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lon Schneider, MD, Study Chair — Keck School of Medicine of USC, Los Angeles, CA
Locations (56):
- United States (56):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Citrials Inc, Bellflower, California
  - Alliance for Research, Long Beach, California
  - Renew Behavioral Health, Inc, Long Beach, California
  - ABS Health LLC, Pomona, California
  - Anderson Clinical Research, Redlands, California
  - Pacific Research Network, Inc, San Diego, California
  - Sharp Mesa Vista Clinical research, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Research Center For Clinical Studies, Inc, Norwalk, Connecticut
  - Pioneer Clinical research, Coconut Creek, Florida
  - University of Miami, Coral Gables, Florida
  - MD Clinical, Hallandale, Florida
  - New Life Medical Research Center, Hialeah, Florida
  - Galiz reserach, Hialeah, Florida
  - Biomed Research Institute, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Advanced Clinical research Network, Miami, Florida
  - Medical Research Group of central Florida Inc., Orange City, Florida
  - The Roskamp Institute, Inc, Sarasota, Florida
  - Infinity Clinical Research, LLC., Sunrise, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Rowe Neurology, Lenexa, Kansas
  - KU School of Medicine-Wichita, Wichita, Kansas
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Pharmasite Research INC, Baltimore, Maryland
  - Quest Research Institute, Farmington Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Galen Research, Chesterfield, Missouri
  - The Neurocognitive Institute, LLC, Mount Arlington, New Jersey
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Global Medical Institutes, Princeton, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Dent Neurosciences Research Center, Inc, Amherst, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New Hope Clinical research, Charlotte, North Carolina
  - Richard H. Weisler, M.D., P.A. & Associates, Raleigh, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Red river medical research Center, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC., Tulsa, Oklahoma
  - The Clinical research Center LLC, Jenkintown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Shepherd Clinical Research LLC, Lewisville, Texas
  - Radiant Research, San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Aspen Clinical research, Orem, Utah
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Zain Research, Llc, Richland, Washington
  - SSM Health/Dean Medical Group, Madison, Wisconsin

REFERENCES:
- [Derived] Schneider LS, Laudon M, Nir T, Caceres J, Ianniciello G, Capulli M, Zisapel N. A Polymorphism Cluster at the 2q12 locus May Predict Response to Piromelatine in Patients with Mild Alzheimer's Disease. J Prev Alzheimers Dis. 2022;9(2):247-254. doi: 10.14283/jpad.2021.61. PMID 35542997
- Available data/document: Study website — http://www.recognitionstudy.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first period of the study consisted of a run-in phase where all participants received Placebo, followed by a second period where participants were randomized to "Piromelatine 5mg", "Piromelatine 20mg", "Piromelatine 50mg", or "Placebo" Arm/Groups for the dose escalation phase.
Groups:
- Experimental: Piromelatine 5 mg: Run-In placebo (2 weeks), followed by 5 mg Piromelatine once daily (26 weeks)
- Experimental: Piromelatine 20 mg: Run-In placebo (2 weeks), followed by 20 mg Piromelatine once daily (26 weeks).
- Experimental: Piromelatine 50 mg: Run-In placebo (2 weeks), followed by 50 mg Piromelatine once daily (26 weeks).
- Placebo Comparator: Run-In placebo (2 weeks), followed by Placebo control once daily (26 weeks).
Period: Run-In Phase (2 Weeks)
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator
Started | 89 | 88 | 88 | 106
Completed | 89 | 88 | 88 | 106
Not Completed | 0 | 0 | 0 | 0
Period: Double Blind Dose Escalation (26 Weeks)
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator
Started | 89 | 88 | 88 | 106
Number of Baseline Participants | 83 | 87 | 80 | 102
Completed | 71 | 88 | 88 | 85
Not Completed | 18 | 0 | 0 | 21

BASELINE CHARACTERISTICS:
Population: Out of 371 patients randomized, 368 were included in the Safety Analysis Set (SS), 352 were in the Full Analysis Set (FAS), and 315 were in the Per Protocol Set (PPS).
  Out of 368 patients included in the SS, 16 were not included in the FAS because they did not have efficacy data for the primary endpoint at baseline and at least 1 postbaseline measurement. Of the 352 patients included in the FAS, 37 patients were not included in the PPS because they experienced major protocol deviations.
Groups:
- Experimental: Piromelatine 5 mg: Piromelatine 5 mg tablet once daily
- Experimental: Piromelatine 20 mg: Piromelatine 20 mg tablet once daily
- Experimental: Piromelatine 50 mg: Piromelatine 50 mg tablet once daily
- Placebo Comparator: Placebo: Placebo tablet given once daily
- Total: Total of all reporting groups
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 83 | 87 | 80 | 102 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 83 | 87 | 80 | 102 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (6.65) | 72.7 (7.97) | 73.3 (6.62) | 73.3 (7.11) | 73.1 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 49 | 49 | 58 | 200
  Male | 39 | 38 | 31 | 44 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 24 | 20 | 83
  Not Hispanic or Latino | 65 | 66 | 56 | 82 | 269
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 11 | 9 | 6 | 8 | 34
  White | 70 | 78 | 72 | 92 | 312
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 87 | 80 | 102 | 352

OUTCOME MEASURES:

1. Primary Outcome: Computerized Neuropsychological Test Battery (cNTB) Z-Scores - Change From Baseline
Description: The global composite score of the cNTB combines the International Shopping List Test (ISLT), One Card Learning (OCL), Identification (IDN), Detection (DET), One Back Card (OBK), Controlled Oral Word Association Test (COWAT), and the Categorical Fluency Test (CFT). For each test, a z-score relative to the study baseline is calculated.
  The cNTB global composite score is the mean of all z-scores from the tests listed above.
  The scale range is from -3 to 3. Zero Z-score means no cognitive change. A negative value means decline, while a positive value means improvement.
Time Frame: 26 weeks
Measure: Mean (95% Confidence Interval); unit: z-score
Groups:
- Piromelatine 5 mg: 5 mg Piromelatine tablets once daily
- Piromelatine 20 mg: 20 mg Piromelatine tablets once daily
- Piromelatine 50 mg: 50 mg Piromelatine tablets once daily
- Placebo Comparator: Placebo tablet once daily
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
z-score | 0.0434 [-0.0728 to 0.1391] | 0.1175 [0.0121 to 0.2153] | 0.0297 [-0.0900 to 0.1247] | 0.0591 [-0.0435 to 0.1483]

2. Secondary Outcome: Change From Baseline in Global Impression of Change (CGIC)
Description: The Change From Baseline in Global Impression of Change (CGIC) rating is made on a 7-point Likert-type scale where the change from baseline is rated as marked improvement (1), moderate improvement (2), minimal improvement (3), no change (4), minimal worsening (5), moderate worsening (6), marked worsening (7).
  Mean values at 13 and 26 weeks are relative to baseline.
Time Frame: 13 weeks, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator: Placebo
Number analyzed (Participants) | 83 | 87 | 80 | 102
score on a scale
  13 weeks | 3.93 (0.88) | 3.95 (0.78) | 3.87 (0.92) | 3.89 (0.80)
  26 weeks | 4.13 (1.07) | 3.94 (1.02) | 3.87 (0.98) | 3.99 (1.01)

3. Secondary Outcome: Alzheimer's Disease Cooperative Study/Activities of Daily Living Scale Adapted for MCI (Mild Cognitive Impairment) Patients (ADCS-MCI-ADL)
Description: ADCS-MCI-ADL is an evaluation scale with information provided by an informant/caregiver to describe the functional impairment of patients with mild cognitive impairment (MCI).
  The ADCS-ADL is a 23-item scale that includes 6 basic ADLs (BADLs) and 17 Instrumental Activities of Daily Living (IADLs) that provide a total score of 0-78, with a lower score indicating greater severity, meaning a worse outcome.
Time Frame: Baseline, 13 weeks, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
score on a scale
  Baseline | 40.7 (6.73) | 38.4 (8.98) | 39.2 (7.60) | 39.4 (8.60)
  13 weeks | 40.4 (6.72) | 39.6 (8.89) | 39.1 (8.81) | 39.5 (8.06)
  26 weeks | 40.6 (6.59) | 39.3 (9.11) | 39.8 (7.94) | 40.4 (8.07)

4. Secondary Outcome: Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-cog14)
Description: The ADAS was designed to measure the severity of the most important symptoms of AD. Its subscale, ADAS-cog, is the most popular cognitive testing instrument used in clinical trials, measuring the disturbances of memory, language, praxis, attention, and other cognitive abilities that are often referred to as the core symptoms of AD.
  ADAS-cog14 comprises 14 items summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment.
Time Frame: Baseline, 13 weeks, and 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Piromelatine 5 mg: 5 mg tablets Piromelatine once daily
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
score on a scale
  Baseline | 26.1 (7.72) | 26.3 (9.16) | 26.4 (7.91) | 26.6 (8.62)
  13 weeks | 25.1 (8.39) | 26.7 (9.37) | 25.5 (10.01) | 26.6 (9.87)
  26 weeks | 25.3 (8.93) | 26.0 (10.12) | 24.9 (9.35) | 25.2 (9.97)

5. Secondary Outcome: Safety and Tolerability - Blood Pressure (mmHg)
Description: Systolic and Diastolic Blood Pressure is followed during the study, as safety and tolerability measures.
  Changes in BP following treatment, leading to values out of the normal limits mean a worse outcome.
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
mmHg
  Systolic BP - Baseline | 128.7 (14.51) | 130.8 (13.19) | 128.5 (11.35) | 132.3 (15.13)
  Systolic BP - 26 weeks | 131.9 (13.61) | 132.4 (12.31) | 129.9 (10.01) | 131.5 (12.93)
  Diastolic BP - Baseline | 75.3 (9.15) | 76.5 (8.37) | 76.3 (7.57) | 76.3 (8.26)
  Diastolic BP - 26 weeeks | 76.3 (8.48) | 76.2 (8.47) | 77.3 (8.78) | 76.3 (8.52)

6. Secondary Outcome: Safety and Tolerability - Heart Rate (Bpm)
Description: Heart Rate within normal limits = 60-100 beats per minute (bpm) during the study means a good outcome in terms of safety.
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator: Placebo
Number analyzed (Participants) | 83 | 87 | 80 | 102
bpm
  Heart rate - baseline | 68.1 (10.67) | 68.7 (9.44) | 69.6 (9.55) | 67.2 (9.68)
  Heart rate - 26 weeks | 65.9 (9.89) | 67.0 (9.95) | 66.9 (9.28) | 67.9 (10.13)

7. Secondary Outcome: Safety and Tolerability - ECG Interval Results - QTcF (Msec)
Description: QT interval corrected for heart rate by Fridericia's cube root formula (QTcF). The QTc is considered normal at < 450 msec in males, and < 470 msec in females.
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator: Placebo
Number analyzed (Participants) | 83 | 87 | 80 | 102
msec
  Baseline | 417.1 (24.16) | 416.4 (34.97) | 413.9 (50.48) | 416.5 (20.57)
  26 weeks | 414.3 (27.29) | 421.2 (24.86) | 416.6 (24.87) | 408.9 (54.47)

8. Secondary Outcome: Safety and Tolerability - Hematology
Description: Hematology (GI/L).
  1 gill (GI) = 0.118294118 liter (L). No major changes or shifts from baseline mean good safety and tolerability.
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
GI/L
  Basophils - baseline | 0.050 (0.0141) | 0.070 (0.0141) | 0.067 (0.0153) | 0.063 (0.0153)
  Basophils - 26 weeks | 0.080 (0) | 0.050 (0) | 0.050 (0.0141) | 0.080 (0.0283)
  Eosinophils - baseline | 0.290 (0.0990) | 0.215 (0.0354) | 0.110 (0.0693) | 0.153 (0.0208)
  Eosinophils - 26 weeks | 0.170 (0) | 0.180 (0) | 0.130 (0.0283) | 0.250 (0.0283)
  Leukocytes - baseline | 6.455 (1.5768) | 8.715 (2.7224) | 6.140 (0.6940) | 5.407 (0.8755)
  Leukocytes - 26 weeks | 5.210 (0) | 10.050 (0) | 5.885 (0.3465) | 6.970 (0.9617)
  Lymphocytes - baseline (GI/L) | 1.605 (0.7425) | 2.535 (0.0071) | 1.943 (0.2397) | 1.363 (0.3320)
  Lymphocytes - 26 weeks | 0.920 (0) | 2.370 (0) | 1.805 (0.3182) | 2.085 (1.3223)
  Monocytes - baseline | 0.510 (0.2828) | 0.405 (0.0919) | 0.357 (0.1102) | 0.347 (0.0611)
  Monocytes - 26 weeks | 0.450 (0) | 0.700 (0) | 0.370 (0.0141) | 0.345 (0.0495)
  Neutrophils - baseline | 3.990 (0.4525) | 5.495 (2.6658) | 3.660 (0.2905) | 3.483 (1.1801)
  Neutrophils - 26 weeks | 3.600 (0) | 6.750 (0) | 3.525 (0.0071) | 4.205 (0.3041)
  Platelets - baseline | 238.5 (84.15) | 299.0 (2.83) | 241.0 (46.13) | 167.3 (26.95)
  Platelets - 26 weeks | 144.0 (0) | 301.0 (0) | 223.0 (48.08) | 283.0 (111.72)

9. Secondary Outcome: Safety and Tolerability - Blood Chemistry (mmol/L)
Description: Blood Chemistry follow-up during the experiment. No major changes or shifts from baseline mean good safety and tolerability.
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Experimental: Piromelatine 5 mg | Experimental: Piromelatine 20 mg | Experimental: Piromelatine 50 mg | Placebo Comparator: Placebo
Number analyzed (Participants) | 83 | 87 | 80 | 102
mmol/L
  Glucose - baseline | 5.89 (1.883) | 5.97 (2.045) | 5.51 (1.322) | 5.78 (1.598)
  Glucose - 26 weeks | 5.86 (1.770) | 6.25 (2.121) | 5.99 (2.351) | 5.80 (1.461)
  Calcium - baseline | 2.385 (0.1626) | 2.470 (0.0707) | 2.307 (0.1007) | 2.363 (0.1290)
  Calcium - 26 weeks | 2.270 (0) | 2.370 (0) | 2.300 (0) | 2.335 (0.0495)
  Sodium - baseline | 140.5 (2.12) | 141.5 (0.71) | 139.3 (2.31) | 139.0 (1.73)
  Sodium -26 weeks | 135.0 (0) | 141.0 (0) | 143.0 (2.83) | 140.0 (1.41)
  Urea Nitrogen - baseline | 7.35 (0.778) | 7.70 (3.818) | 5.00 (0.400) | 5.00 (1.212)
  Urea Nitrogen - 26 weeks | 8.20 (0) | 5.70 (0) | 5.35 (0.495) | 4.50 (1.273)

10. Other Pre Specified Outcome: NeuroPsychiatric Inventory (NPI) Total Score
Description: The NPI scale consists of 12 domains that are rated for both frequency (range 1 to 4) and severity (range 1 to 3). A composite score for each domain is calculated (frequency × severity), and it ranges from 1 to 12.
  For each item, there is a leading question. If the symptom is absent, then the frequency, severity, and distress scores are not completed. In this case, the score is 0 for the item. The sum of the composite scores yields the NPI total score (1-12).
  A negative change in the score indicates an improvement from baseline (symptom reduction).
Time Frame: Baseline, and 26 weeks
Measure: Mean (Standard Deviation); unit: NPI total score
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
NPI total score
  Baseline | 11.2 (10.30) | 10.3 (8.39) | 12.0 (8.75) | 10.8 (10.13)
  26 weeks | 11.4 (11.60) | 9.0 (7.85) | 11.9 (10.66) | 9.8 (10.34)

11. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (PSQI) - Global Component Score
Description: PSQI is an effective instrument used to measure the quality and patterns of sleep in older adults.
  It differentiates "poor" from "good" sleep by measuring 7 areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month.
  PSQI includes seven components, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: Baseline, 4 weeks, 13 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: PSQI global score
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator
Number analyzed (Participants) | 83 | 87 | 80 | 102
PSQI global score
  Baseline | 6.8 (4.39) | 5.9 (3.99) | 6.0 (4.14) | 5.6 (3.66)
  4 weeks | 5.8 (3.97) | 5.4 (3.36) | 5.4 (3.56) | 5.6 (3.39)
  13 weeks | 6.2 (3.85) | 5.2 (3.04) | 5.5 (3.20) | 5.1 (3.11)
  26 weeks | 5.7 (3.62) | 4.7 (3.26) | 5.2 (3.21) | 5.1 (3.68)

ADVERSE EVENTS:
Time Frame: 28 weeks (2 weeks Run-In Phase + 26 weeks Dose Escalation Phase)
Description: The data presented includes adverse events from the Run-In Phase (2 weeks of placebo, intended to assess eligibility into the dose escalation study), and the Dose Escalation Phase (26 weeks of treatment with investigational drug versus placebo).
Groups:
- Piromelatine 5 mg: 5 mg Piromelatine tablets once daily for 26 weeks (Dose Escalation Phase = Weeks 2-28).
- Piromelatine 20 mg: 20 mg Piromelatine tablets once daily for 26 weeks (Dose Escalation Phase = Weeks 2-28).
- Piromelatine 50 mg: 50 mg Piromelatine tablets once daily for 26 weeks (Dose Escalation Phase = Weeks 2-28).
- Placebo Comparator: Placebo tablet once daily for 26 weeks (Dose Escalation Phase = Weeks 2-28).
- Run-In Phase: Placebo tablet once daily for 2 weeks, intended to assess eligibility before starting the dose escalation phase (Weeks 0-2).
Arm/Group | Piromelatine 5 mg | Piromelatine 20 mg | Piromelatine 50 mg | Placebo Comparator | Run-In Phase
All-Cause Mortality (participants affected / at risk) | 1/88 | 0/88 | 0/87 | 0/105 | 0/368
Serious Adverse Events (participants affected / at risk) | 2/88 | 6/88 | 4/87 | 6/105 | 0/368
Other Adverse Events (participants affected / at risk) | 12/88 | 14/88 | 14/87 | 29/105 | 0/368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Piromelatine 5 mg (N=88) | Piromelatine 20 mg (N=88) | Piromelatine 50 mg (N=87) | Placebo Comparator (N=105) | Run-In Phase (N=368)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) — Pneumonia
Kidney Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Kidney Infection
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Head Injury
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Fall
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Ischaemic cardiomyopathy
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subdural haematoma
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Malignant melanoma in situMalignant melanoma in situ
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Duodenal ulcer
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Duodenitis
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Gastritis erosive
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Gastrointestinal haemorrhage
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory failure
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Colitis
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cervix carcinoma
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Uterine cancer
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Acute myocardial infarction
Femur Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Femur Fracture
Humerus Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Humerus Fracture
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Bradycardia
Cardio-respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Cardio-respiratory Arrest
Ischemic Cardiopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Ischemic Cardiopathy
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Squamous cell carcinoma of skin
Syncope (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Syncope
Transient ischaemic attack (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Transient ischaemic attack
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Anaemia
Multi-organ disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Multi-organ disorder
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Anxiety
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Piromelatine 5 mg (N=88) | Piromelatine 20 mg (N=88) | Piromelatine 50 mg (N=87) | Placebo Comparator (N=105) | Run-In Phase (N=368)
Headache (Nervous system disorders) | 0 (0) | 3 (6) | 1 (1) | 8 (15) | 0 (0) — Headache
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) — Abnormal dreams
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) — Dizziness
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Somnolence
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Head discomfort
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hypersomnia
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Sedation
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Insomnia
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Agitation
Initial insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Initial insomnia
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Disorientation
Disturbance in sexual arousal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Disturbance in sexual arousal
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hallucination
Libido increased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Libido increased
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (5) | 0 (0) — Nausea
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) — Constipation
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Diarrhoea
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Large intestine polyp
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Abdominal distension
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Abdominal pain
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dry mouth
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dyspepsia
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Gastrooesophageal reflux
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) — Nasopharyngitis
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Kidney infection
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Sinusitis
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Upper respiratory tract infection
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Influenza
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Staphylococcal infection
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Tubo-ovarian abscess
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Alopecia
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dry skin
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Rash
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Fall
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Cough
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dyspnoea
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Oropharyngeal pain
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Asthenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT02615002/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT02615002/SAP_001.pdf